CLINICAL TRIAL: NCT02244892
Title: Correlation of Scheimpflug Densitometry Measurements of Corneal Haze With Disability Glare
Status: Withdrawn | Type: Observational
Why Stopped: Recruitment
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 04-14-30
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Vision Disability
Keywords: Disability glare; Corneal scar; Corneal haze; Scheimpflug densitometry; Contrast sensitivity
MeSH Terms: conditions — Vision Disorders; Corneal Injuries; Corneal Opacity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Disability glare is described as "halos" or "starbursts" around bright sources of light that can cause discomfort and reduce vision. The cornea is the clear "window" at the front of the eye, but certain conditions such as a previous infection can leave a scar. Corneal scars can cause disability glare by scattering and spreading incoming light instead of allowing it to focus on the back of the eye (retina) to get a crisp image. In this study, the corneal scar will be analyzed using a new device that measures scar density (Pentacam), and a relationship with disability glare will be made. This can help us further understand disability glare and make better decisions in the future on when to treat these scars to help patients see better.

DETAILED DESCRIPTION:
Disability glare is a phenomenon commonly described as starbursts and halos that results in difficulty seeing clearly in the presence of bright "blinding" light. It can appear as if a veil of light is cast over the world outside. Optically, this occurs when incoming light is scattered in the eye instead of being focused on the retina. This is called straylight, and it diffusely illuminates the retina which causes desensitization of the photoreceptors and reduces the contrast of the retinal image (Lombardo & Lombardo, 2010). The main sources of scatter in the human eye are opacities in the clear ocular media, primarily due to diffusion and loss of transparency in the cornea and lens, as well as within the retina. While the lens is the largest contributor to light scatter (especially with cataract formation and aging), opacification of the cornea (e.g. scars or haze) can similarly cause intraocular light scattering, resulting in disability glare and decreased contrast sensitivity (Fan-Paul et al., 2002).

Due to the subjective nature of disability glare and contrast sensitivity, it is fairly difficult to develop a reliable objective way to measure and quantify this phenomenon. One of the most commonly used clinical tests for disability glare is the Brightness Acuity Tester (BAT), which is described as an ice cream scooper 60 mm in diameter with a 12 mm hole in the center. With the patient viewing a visual acuity chart through the hole, a uniform luminance at three different settings-high (white sand beach), medium (clear day), low (overhead lighting)-is used to induce glare and simulate the various real-life conditions. The drop in visual acuity with the various glare settings is used as a measure of disability glare. The BAT test has been found to be a reliable predictor of outdoor visual acuity (clinically validated for use in measuring disability glare secondary to cataracts), is ubiquitously available, and is easy to administer. To further and more accurately reflect real life situations, it can be used in conjunction with a contrast sensitivity chart rather than the regular black-on-white Snellen letter chart (Aslam et al., 2007). Contrast sensitivity can be tested using letter-based charts (e.g. Pelli-Robson letter sensitivity chart) that consist of letters of the same size but with decreasing contrast, or contrast gratings, which are based on sinusoidal waves of light (e.g. Vistech MCT-8000 or FACT).

Opacification of the cornea in the form of scars or haze is a natural response to a wide array of pathological insults (e.g. infection, degeneration, corneal dystrophies) and can result in light scatter and glare. Measurement of corneal haze was previously crudely performed via standard slit-lamp examination and human measurement. Recently, an automated, non-invasive, and objective method to measure corneal scar density was introduced using Scheimpflug imaging. This Pentacam device (Oculus Optikgerate GmbH, Wetzlar, Germany) consists of a rotating camera that captures images of the cornea at an angle, and analysis of these anterior segment images can be employed to quantify scattered light in various diameters and depths of the cornea. The generated maps of the amount of scatter in different regions of the cornea are called corneal densitometry maps, and they are displayed along with maps of corneal topography (elevation) and pachymetry (thickness). Normative values for Scheimpflug densitometry have recently been established (Dhubhghaill et al., 2013). Measurements have also been obtained after various surgical procedures to analyze their impact on corneal clarity. This includes analysis of corneas after refractive surgery such as LASIK (Cennamo et al., 2011; Fares et al., 2012) and PRK (Takacs et al., 2011), as well as various forms of corneal transplantation (Koh et al., 2012; Bhatt et al., 2012; Arnalich-Montiel et al., 2013; Ivarsen & Hjortdal, 2013) and collagen cross-linking (Gutierrez et al., 2012; Greenstein et al., 2010). Furthermore, it has been used to characterize pathological conditions including infectious keratitis (Otri et al., 2012; Orucoglu et al., 2014) and congenital corneal opacities (Elfein et al., 2013). However, no functional correlation has been made with these anatomical maps, and the relationship between scattered light as measured by densitometry and its effect on visual function such as contrast sensitivity and disability glare has not been well-characterized.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Presence of corneal scar in one eye
* No clinical evidence of any other intraocular pathology

Exclusion Criteria:

* Clinical evidence of other ocular pathology (e.g. cataracts)
* Pediatric patients less than 18 years old
* Bilateral corneal pathology
* Presence of active corneal inflammation/infection
* Presence of degenerative corneal disease
* History of prior corneal surgery (e.g. corneal graft)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective study in which all eligible and willing patients will undergo the same workup. The expected duration is 1 year, and the trial will be stopped once the needed number of subjects has been enrolled. Testing will be performed on the day of the routine clinical visit and will only extend the appointment by less than 30 minutes.
  All patients receiving ophthalmological care at University Hospitals (both at the main Case Medical Center site and the satellite offices at Westlake and Landerbrook) who meet the inclusion and exclusion criteria would be eligible for this study. Subjects will be identified who have an isolated corneal scar in one eye and otherwise healthy eyes with no clinical evidence of lens or retinal pathology. Patients will be enrolled between September 6, 2014 and September 5, 2015, with the goal of recruiting at least 80-100 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Disability glare | 1 year
  BAT measurements of disability glare
Visual quality | 1 year
  NEI-VFQ25 questionnaire on functional visual quality
Contrast sensitivity | 1 year
  Vistech contrast grating test
Visual acuity | 1 year
  Visual acuity measured by Snellen chart

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Fan-Paul NI, Li J, Miller JS, Florakis GJ. Night vision disturbances after corneal refractive surgery. Surv Ophthalmol. 2002 Nov-Dec;47(6):533-46. doi: 10.1016/s0039-6257(02)00350-8. PMID 12504738
- [Background] Aslam TM, Haider D, Murray IJ. Principles of disability glare measurement: an ophthalmological perspective. Acta Ophthalmol Scand. 2007 Jun;85(4):354-60. doi: 10.1111/j.1600-0420.2006.00860.x. Epub 2007 Feb 20. PMID 17313443
- [Background] Lombardo M, Lombardo G. Wave aberration of human eyes and new descriptors of image optical quality and visual performance. J Cataract Refract Surg. 2010 Feb;36(2):313-31. doi: 10.1016/j.jcrs.2009.09.026. PMID 20152616
- [Background] Ni Dhubhghaill S, Rozema JJ, Jongenelen S, Ruiz Hidalgo I, Zakaria N, Tassignon MJ. Normative values for corneal densitometry analysis by Scheimpflug optical assessment. Invest Ophthalmol Vis Sci. 2014 Jan 7;55(1):162-8. doi: 10.1167/iovs.13-13236. PMID 24327608
- [Background] Cennamo G, Forte R, Aufiero B, La Rana A. Computerized Scheimpflug densitometry as a measure of corneal optical density after excimer laser refractive surgery in myopic eyes. J Cataract Refract Surg. 2011 Aug;37(8):1502-6. doi: 10.1016/j.jcrs.2011.03.037. PMID 21782093
- [Background] Fares U, Otri AM, Al-Aqaba MA, Faraj L, Dua HS. Wavefront-optimized excimer laser in situ keratomileusis for myopia and myopic astigmatism: refractive outcomes and corneal densitometry. J Cataract Refract Surg. 2012 Dec;38(12):2131-8. doi: 10.1016/j.jcrs.2012.07.041. Epub 2012 Oct 18. PMID 23084157
- [Background] Takacs AI, Mihaltz K, Nagy ZZ. Corneal density with the Pentacam after photorefractive keratectomy. J Refract Surg. 2011 Apr;27(4):269-77. doi: 10.3928/1081597X-20100618-02. Epub 2010 Jul 1. PMID 20672772
- [Background] Koh S, Maeda N, Nakagawa T, Nishida K. Quality of vision in eyes after selective lamellar keratoplasty. Cornea. 2012 Nov;31 Suppl 1:S45-9. doi: 10.1097/ICO.0b013e318269c9cd. PMID 23038035
- [Background] Bhatt UK, Fares U, Rahman I, Said DG, Maharajan SV, Dua HS. Outcomes of deep anterior lamellar keratoplasty following successful and failed 'big bubble'. Br J Ophthalmol. 2012 Apr;96(4):564-9. doi: 10.1136/bjophthalmol-2011-300214. Epub 2011 Dec 1. PMID 22133987
- [Background] Arnalich-Montiel F, Hernandez-Verdejo JL, Oblanca N, Munoz-Negrete FJ, De Miguel MP. Comparison of corneal haze and visual outcome in primary DSAEK versus DSAEK following failed DMEK. Graefes Arch Clin Exp Ophthalmol. 2013 Nov;251(11):2575-84. doi: 10.1007/s00417-013-2460-y. Epub 2013 Sep 6. PMID 24008847
- [Background] Ivarsen A, Hjortdal J. Recipient corneal thickness and visual outcome after Descemet's stripping automated endothelial keratoplasty. Br J Ophthalmol. 2014 Jan;98(1):30-4. doi: 10.1136/bjophthalmol-2013-304042. Epub 2013 Oct 16. PMID 24133026
- [Background] Gutierrez R, Lopez I, Villa-Collar C, Gonzalez-Meijome JM. Corneal transparency after cross-linking for keratoconus: 1-year follow-up. J Refract Surg. 2012 Nov;28(11):781-6. doi: 10.3928/1081597X-20121011-06. PMID 23347372
- [Background] Greenstein SA, Fry KL, Bhatt J, Hersh PS. Natural history of corneal haze after collagen crosslinking for keratoconus and corneal ectasia: Scheimpflug and biomicroscopic analysis. J Cataract Refract Surg. 2010 Dec;36(12):2105-14. doi: 10.1016/j.jcrs.2010.06.067. PMID 21111314
- [Background] Otri AM, Fares U, Al-Aqaba MA, Dua HS. Corneal densitometry as an indicator of corneal health. Ophthalmology. 2012 Mar;119(3):501-8. doi: 10.1016/j.ophtha.2011.08.024. Epub 2011 Nov 30. PMID 22133793
- [Background] Elflein HM, Hofherr T, Berisha-Ramadani F, Weyer V, Lampe C, Beck M, Pitz S. Measuring corneal clouding in patients suffering from mucopolysaccharidosis with the Pentacam densitometry programme. Br J Ophthalmol. 2013 Jul;97(7):829-33. doi: 10.1136/bjophthalmol-2012-302913. Epub 2013 May 17. PMID 23685998